CLINICAL TRIAL: NCT05914194
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate the Efficacy and Safety of NLS-2 (Mazindol Extended-Release) Tablets in the Treatment of Narcolepsy Type 1
Brief Title: A Eight-Week Study of NLS-2 (Mazindol Extended Release) in Participants With Narcolepsy Type 1
Acronym: AMAZE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NLS Pharmaceutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NLS-1031
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Narcolepsy Type 1; Narcolepsy With Cataplexy
Keywords: Narcolepsy; Cataplexy; Narcolepsy Type 1; Narcolepsy with Cataplexy
MeSH Terms: conditions — Narcolepsy; Cataplexy

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NLS-2 (Experimental): Participants will receive a single NLS-2 tablet orally once daily from Day 1 to Day 56 (until the end of Week 8).
  Interventions: Drug: NLS-2
- Placebo (Placebo Comparator): Participants will receive a single NLS-2 placebo matching tablet orally once daily from Day 1 to Day 56 (until the end of Week 8).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NLS-2 — Participants will receive NLS-2 tablets orally.
  Other Names: mazindol extended-release (ER), mazindol controlled-release (CR)
  Arms: NLS-2
Drug: Placebo — Participants will receive NLS-2 matching placebo tablets orally.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to see how NLS-2 (mazindol extended-release) works on symptoms of narcolepsy, including cataplexy and excessive daytime sleepiness.

Approximately 48 participants will take part in the study across the United States.

The study treatment (NLS-2 or placebo) will be administered for 8 weeks. After this treatment period, the participant may have the option to participate in a separate long-term extension study during which all participants will be treated with NLS-2.

DETAILED DESCRIPTION:
This is a Phase 3, double-blind, placebo-controlled, multicenter, randomized, parallel-group clinical trial. The primary goal of this study is to assess the efficacy and safety of NLS-2 (mazindol extended-release) tablets in treating Narcolepsy Type 1. The trial aims to determine the effects of NLS-2 on the improvement of narcolepsy symptoms, including cataplexy frequency and excessive daytime sleepiness.

Participants in this trial will receive either NLS-2 or a placebo for 8 weeks. The treatment assignment will be concealed from both the participant and the investigator throughout the trial (unless there is an urgent medical need).

Approximately 48 patients will be enrolled at multiple clinical sites across the United States. Following the completion of the trial, participants may be given the option to enroll in a separate long-term extension trial where all participants will receive NLS-2 treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥ 18 years of age at the time of signing the informed consent.
* Documented primary diagnosis of Narcolepsy Type 1 (NT1) according to the International Classification of Sleep Disorders-Third Edition (ICSD-3) criteria.
* Willing and able to safely discontinue all prohibited medications, including medications for the treatment of narcolepsy.
* Body Mass Index (BMI) within the range of 18 - 40 kg/m2 (inclusive).

Key Exclusion Criteria:

* Any other (besides narcolepsy) clinically relevant medical, behavioral, or psychiatric disorder that is associated with excessive daytime sleepiness or cataplexy.
* History of myocardial infarction or significant cardiovascular disease, structural cardiac abnormalities, cardiomyopathy, congestive heart failure, cardiac arrhythmias, coronary artery disease, cerebrovascular disease (transient ischemic attack or stroke), or any other significant cardiac problem.
* History of long QT Syndrome or Torsades de Pointes, or an immediate family history of sudden cardiac death.
* History of pulmonary hypertension and/or valvulopathy.
* History of epilepsy, convulsions, or seizures (excluding early childhood febrile seizures).
* Significant history of head injury or head trauma.
* Recent or active suicidal ideation or behavior
* Current, or within the past year, diagnosis of substance abuse or dependence disorder (SUD) including alcohol abuse.
* Narrow-angle glaucoma.
* Severe renal or hepatic insufficiency.
* Occupation that requires variable or nighttime shift work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of cataplexy episodes at Week 8 | 8 weeks
  Cataplexy episodes is a clinical outcome measure that assesses the frequency of cataplexy episodes.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System-Sleep Related Impairment (PROMIS-SRI): change from baseline | 8 weeks
  The Patient Reported Outcomes Measurement Information System-Sleep Related Impairment (PROMIS-SRI) scale consists of 8 items to evaluate daytime consequences of functioning on a 5-point Likert scale ranging from 1 to 5. The PROMIS-SRI measures self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Each question has five response options ranging in value from 1 to 5. To find the total raw score with all questions answered, sum the values of the response to each question and total score ranges from 8 to 40. Higher scores indicates greater sleep impairment.
Patient Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD): change from baseline | 8 weeks
  The Patient Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) consists of a static 8-item questionnaire. Using a recall period of the past 7 days, it assesses the concepts of sleep initiation (2 items), quality of sleep (3 items), early morning feelings (2 items) and worrying about sleep (1 item). Each question has 5 response options ranging in value from 1 to 5. To find the total raw score with all questions answered, sum the values of the response to each question and a total score ranges from 8 to 40. Lower scores indicate less sleep disturbance. Negative changes in scores indicate improvement.
Epworth Sleepiness Scale (ESS): change from baseline | 8 weeks
  The Epworth Sleepiness Scale (ESS) is a patient-reported outcome measure that assesses daytime sleepiness. It asks the participant to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep in 8 different situations or activities that are commonly met in daily life. The total ESS score, ranging from 0 to 24, is the sum of 8 item scores, with higher scores indicating greater daytime sleepiness.
Patient Global Impression of Severity (PGI-S): change from baseline | 8 weeks
  The Patient Global Impression of Severity (PGI-S) is a patient-reported outcome measure that assesses the participant's perception of the severity of their illness. The participant rates their condition on a point scale, from "no symptoms" to "extremely severe."
Clinician Global Impression of Severity (CGI-S): change from baseline | 8 weeks
  The Clinical Global Impressions of Severity (CGI-S) is a clinician-rated outcome measure that assesses the clinician's impression of the participant's current illness severity. The clinician rates the severity of the participant's condition on a point scale, from "normal, not at all ill" to "among the most extremely ill patients".

CONTACTS AND LOCATIONS:
Overall Officials: George Apostol, MD, MS, Study Chair — NLS Pharmaceutics

IPD SHARING:
Plan to Share IPD: No